CLINICAL TRIAL: NCT02566668
Title: Immune Airway-Epithelial Interactions in Steroid-Refractory Severe Asthma
Brief Title: Immune Interactions in Severe Asthma
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sally E. Wenzel MD, MD, University of Pittsburgh
Other Study IDs: PRO15050456
Record Dates: First submitted 2015-09-18; First posted 2015-10-02 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: Asthma; Severe Asthma; IL-10; IL-27; IL-13; Epithelial Cells; T lymphocytes; Interferon-g
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood - total and specific Immunoglobulin E (IgE); complete blood count; plasma and serum; Deoxyribonucleic Acid (DNA); peripheral blood mononuclear cells (PBMC) Endobronchial biopsy Endobronchial brushings Pulmonary Lavage Exhaled Breath Condensate (EBC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthmatic: 1 year observational follow-up
  Interventions: Other: 1 year Observational Follow-up
- Non-Asthmatic: 1 year observational follow-up
  Interventions: Other: 1 year Observational Follow-up

INTERVENTIONS:
Other: 1 year Observational Follow-up — Approximately 12 months after research bronchoscopy, subjects will return for follow-up visit.

SUMMARY:
This research study is being done to learn more about severe asthma by comparing people with severe asthma to those with milder forms of asthma and people without asthma, at baseline and over time. Individuals are being asked to join a research study to help understand the differences in the lungs and blood of participants with severe asthma compared to those with milder asthma and healthy individuals, as well as differences in overall health. Investigators also want to determine whether these differences predict asthma-related and biologic outcomes over 1 year of follow up.

DETAILED DESCRIPTION:
This study will obtain human lung samples by bronchoscopy from a range of asthmatics and healthy controls to address questions related to the mechanisms for the development of the complex immune processes observed in the lungs. Samples will be evaluated for Type-1, Type-2 and Interleukin-27 (IL-27) expression (and their downstream signatures). In addition, these samples will be evaluated for the presence or absence of Interleukin-10 (IL-10) as a counter regulatory pathway. These pathways will be directly evaluated in epithelial brushings and bronchoalveolar lavage (BAL) cells, as well as BAL fluid. Broad gene expression profiling (Ribonucleic acid (RNA)-sequencing) will also be performed to determine the range of immune-inflammatory markers present in these severe asthmatics. Investigators will specifically address the Signal Transducers and Activators of Transcription (STAT) signaling pathways, particularly STAT-1 and STAT-3 to determine the pattern of activation and downstream responses to develop new therapies. Additionally, in a subset, investigators will compare targeted and untargeted gene expression as obtained from bronchoscopic samples with expression obtained from clinically performed video assisted thoracoscopic (VATS) biopsies of very severe systemic corticosteroid dependent patients. The ultimate goal of this studies is to determine whether a predictive biomarker panel can be identified in the less invasive bronchoscopic samples which predict the findings seen on VATS biopsy.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Non-smoker
* Asthmatic subjects must also demonstrate forced expiratory volume in 1 second (FEV1) bronchodilator reversibility ≥12% or airway hyperresponsiveness reflected by a methacholine provocative concentration causing a 20% fall in FEV1 (PC20) ≤16 mg/mL (Historical methacholine data from previous National Institutes of Health (NIH) trial will be allowed)

Exclusion Criteria:

* Greater than 10 pack year smoking history (none in the last year)
* Vocal cord dysfunction, cystic fibrosis or chronic obstructive pulmonary disorder
* Other lung disease, or any coronary artery disease, hypertension, diabetes or renal failure that is not well-controlled.

Healthy Controls only: Pre-bronchodilator FEV1/Forced vital capacity (FVC) <0.70 or an improvement in FEV1 of more than 12% following 4 puffs of albuterol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected using a Research Registry and clinic patients of the Investigators.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Eotaxin-3 and IL-27 expression and their downstream signatures | 1 Year
  Measure eotaxin-3 and IL-27 expression in bronchoalveolar lavage cells and epithelial cells.

SECONDARY OUTCOMES:
Global gene expression in the airway epithelium and bronchoalveolar lavage cells using RNA-sequencing | 1 Year
Signal transducer and activator of transcription (STAT) signaling pathways | 1 Year
  Pattern of activation and downstream responses
Targeted and untargeted gene expression as obtained from bronchoscopic samples | 1 Year
  Compare with expression obtained from video assisted thoracoscopic (VATS) biopsies of systemic corticosteroid dependent patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sally E Wenzel, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Asthma Institute at UPMC, Pittsburgh, Pennsylvania, United States